CLINICAL TRIAL: NCT05134597
Title: Th17- Gene Expression Profile in Patients With Chronic Venous Leg Insufficiency and Ulcers: Genetical and Clinical Outcomes
Brief Title: Gene Expression in Chronic Venous Leg Ulcers
Acronym: GECVELUS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Catanzaro (Other)
Responsible Party: Principal Investigator, Prof. Raffaele Serra, MD, Ph.D., Associate Professor of Vascular Surgery, University of Catanzaro
Other Study IDs: E.R.ALL.2018.42
Record Dates: First submitted 2021-11-14; First posted 2021-11-26 (Actual); Last update posted 2021-11-26 (Actual); Status verified 2021-11

CONDITIONS: Genetic Predisposition to Disease; Inflammation; Venous Leg Ulcer
MeSH Terms: conditions — Genetic Predisposition to Disease; Inflammation; Varicose Ulcer

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1 - Patients with Chronic Venous Disease (CVD): Patients with CVD at different stages, according to CEAP Classification of Chronic Venous Disorders, will be recruited.
  Interventions: Genetic: Genetic assessment
- Group 2 - Healthy subjects without Chronic Venous Disease (CVD): Voluntary healthy subjects without Chronic Venous Disease (CVD) will be recruited.
  Interventions: Genetic: Genetic assessment

INTERVENTIONS:
Genetic: Genetic assessment — Blood samples will be collected in 3-mL K3 EDTA vacutainer tubes. Peripheral blood mononuclear cells will be isolated via density gradient centrifugation within 2 hours of sample collection. Primary CD4+ T cells will be purified from the peripheral blood lymphocytes using a magnetic cell sorting CD4+ T cell isolation kit, according to the manufacturer's instructions. RNA extraction will be performed. Total RNA will be quantified, and the quality of RNA will be assayed using formaldehyde agarose gel electrophoresis and by determining the 260/280 absorbance ratio. One microgram of total RNA from each sample will be subjected to reverse transcription. One microliter of cDNA will be amplified via real-time PCR and 10 pmol of primers specific to IL23R, IL17, SGK1, RANBP1, TFGB. Real-time PCR assays will be performed in triplicate The specificity of the PCR products will be determined via melting curve analysis.

SUMMARY:
Chronic Venous Disease (CVD) is a widespread clinical condition widely spread in the western countries that may negatively impact the quality of life (QoL) of affected patients. Chronic venous leg ulcers (CVLUs) are the most severe form of CVD, and several genetic and molecular alterations have been studied in order to understand the progression of CVD towards CLVUs. Chronic inflammation is a key element in CVLUs onset, and recently T helper 17 (Th-17) cells, a subtype of pro-inflammatory T helper (CD4+) cells defined by the production of a cytokine signature of which IL-17 represents the progenitor, seem to be related to several chronic disease. The aim of this study is to evaluate Th17- Gene Expression profile in patients with CVD and CVLUs.

DETAILED DESCRIPTION:
Chronic Venous Disease (CVD) is a widespread clinical condition widely spread in the western countries, with a prevalence ranging from 10% in adults younger than 30 years of age to nearly 80% for individuals >70 years of age. CVD clinical manifestations vary from mild clinical signs, including varicose veins, to more advanced and severe signs such as chronic venous leg ulcers (CVLUs) which significantly impact the quality of life (QoL) of affected patients. Several genetic and molecular alterations have been studied so far to understand the onset, progression, and complications of CVD, including Chronic Venous Insufficiency (CVI) states in which CVLUs may develop. The appearance of CVLUs is generally preceded by skin changes of the lower limbs such as lipodermatosclerosis, that is a chronic inflammatory condition due to CVI, characterised by an inflammatory skin condition. This pathological event leads to subcutaneous fibrosis and hardening of the affected skin, resulting in tissue hypoxia essential for venous ulceration.Gene expression profile studies, present in the current literature, allow us to hypothesize several mechanisms underlying the development of CVLU, highlighting a wide variety of genetic-molecular interconnections. Nevertheless, none to date is able to provide a genetic and cellular model linking the pathogenetic events that lead to the onset of CVLU or the progression of these lesions.T helper 17 (Th-17) cells are a subtype of pro-inflammatory T helper (CD4+) cells defined by the production of a cytokine signature of which IL-17 represents the progenitor. The development and differentiation and expansion of Th-17 depends on differentiation factors (TGF- β ), growth factors (IL-23/IL23R) and several transcription factors (ROR-γt, STAT3 ).

Interestingly, the Th-17 axis has been implicated in several autoimmune diseases including rheumatoid arthritis, multiple sclerosis, ulcerative colitis, Crohn's disease, psoriasis, and autoimmune encephalitis among others. In addition, an increasingly strong role of the Th-17 axis in tumor drug resistance and in the progression and radicalization of HIV infection is recently emerging.

Our study aims at evaluation Th17- Gene Expression profile in patients with CVD and CVLUs.

ELIGIBILITY:
Inclusion Criteria:

* patients with chronic venous disease with CEAP Clinical classes (C) 2-6: C2: varicose veins C3: edema C4: skin changes C5: healed venous ulcers C6: active venous ulcers

Exclusion Criteria:

* patients with peripheral artery disease
* patients with malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with chronic venous disease according to CEAP Classification of Chronic Venous Disorders with clinical classes 2-6.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
Th17- Gene Expression profile | 1 year
  Genetic profile in patients with Chronic Venous Disease and in Healthy subjects will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Raffaele Serra, M.D., Ph.D., Study Chair — University Magna Graecia of Catanzaro
Locations (1):
- University Magna Graecia of Catanzaro, Catanzaro, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Serra R, Ssempijja L, Provenzano M, Andreucci M. Genetic biomarkers in chronic venous disease. Biomark Med. 2020 Feb;14(2):75-80. doi: 10.2217/bmm-2019-0408. Epub 2020 Feb 13. No abstract available. PMID 32053001
- [Background] Metzinger L, de Franciscis S, Serra R. The Management of Cardiovascular Risk through Epigenetic Biomarkers. Biomed Res Int. 2017;2017:9158572. doi: 10.1155/2017/9158572. Epub 2017 Jul 13. PMID 28785591
- [Background] de Franciscis S, Metzinger L, Serra R. The Discovery of Novel Genomic, Transcriptomic, and Proteomic Biomarkers in Cardiovascular and Peripheral Vascular Disease: The State of the Art. Biomed Res Int. 2016;2016:7829174. doi: 10.1155/2016/7829174. Epub 2016 May 19. PMID 27298828
- [Background] Serra R, Buffone G, de Franciscis A, Mastrangelo D, Molinari V, Montemurro R, de Franciscis S. A genetic study of chronic venous insufficiency. Ann Vasc Surg. 2012 Jul;26(5):636-42. doi: 10.1016/j.avsg.2011.11.036. PMID 22664280
- [Background] Kim JS, Jordan MS. Diversity of IL-17-producing T lymphocytes. Cell Mol Life Sci. 2013 Jul;70(13):2271-90. doi: 10.1007/s00018-012-1163-6. Epub 2012 Oct 4. PMID 23052209
- [Background] Smith PD. Update on chronic-venous-insufficiency-induced inflammatory processes. Angiology. 2001 Aug;52 Suppl 1:S35-42. doi: 10.1177/0003319701052001s05. PMID 11510595
- [Background] Moseley TA, Haudenschild DR, Rose L, Reddi AH. Interleukin-17 family and IL-17 receptors. Cytokine Growth Factor Rev. 2003 Apr;14(2):155-74. doi: 10.1016/s1359-6101(03)00002-9. PMID 12651226
- [Derived] Amato R, Dattilo V, Brescia C, D'Antona L, Iuliano R, Trapasso F, Perrotti N, Costa D, Ielapi N, Aiello F, Provenzano M, Bracale UM, Andreucci M, Serra R. Th17-Gene Expression Profile in Patients with Chronic Venous Disease and Venous Ulcers: Genetic Modulations and Preliminary Clinical Evidence. Biomolecules. 2022 Jun 28;12(7):902. doi: 10.3390/biom12070902. PMID 35883458